CLINICAL TRIAL: NCT00330850
Title: An Efficacy Study of a Single Dose Treatment of PRO-513 for Subjects Suffering a Migraine Attack
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ProEthic Pharmaceuticals (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-513301
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2007-04-02 (Estimated); Status verified 2007-03

CONDITIONS: Migraine; Photophobia; Phonophobia
Keywords: Migraine; Photophobia; Phonophobia; Aura
MeSH Terms: conditions — Migraine Disorders; Photophobia; Hyperacusis; Epilepsy | interventions — Diclofenac

INTERVENTIONS:
Drug: PRO-513

SUMMARY:
The purpose of the study is to show the efficacy of a single dose of PRO-513 for treating subjects suffering moderate pain form a migraine attack, with or without aura. The study is also intended to show the effectiveness of PRO-513 for associated symptoms of nausea, photophobia, and phonophobia due to a migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects
* 18-65 years of age
* Primary diagnosis of migraine attack with aura or migraine attack without aura
* Migraine history of averaging at least 1 migraine attack per month but averaging not more than 6 migraine attacks per month over the prior year
* Female subjects must use an effective form of birth control
* Listing of additional inclusion criteria are available through the Sponsor

Exclusion Criteria:

* Excluding subjects with a history of other serious events causing secondary headaches
* Excluding subjects with a current medical condition that could interfere with the overall study intent or affect the absorption, distribution, metabolism, or excretion of the study medication
* Excluding subjects with a history or current medical condition that could confound the study results or use of a concomitant medication that could interfere with the study drug
* Listing of additional exclusion criteria are available through the Sponsor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2006-05; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lipton, MD, Principal Investigator — Montefiore Headache Center
Locations (16):
- United States (16):
  - Associated Neurologists of Southern CT, Fairfield, Connecticut
  - New England Center for Headache, Stamford, Connecticut
  - LCFP Inc., Fort Myers, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - International Research Center, Towson, Maryland
  - Michigan Head-Pain and Neurologic Institute, Ann Arbor, Michigan
  - Mercy Health Research, St Louis, Missouri
  - New York Headache Center, New York, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc., Bryan, Texas
  - Houston Headache Clinic, Houston, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - The Innovative Clinical Research Center, Alexandria, Virginia
  - Advanced Healthcare, S.C., Milwaukee, Wisconsin